CLINICAL TRIAL: NCT05463276
Title: The Characteristics and Risk Factors of Breast Cancer Patients Trend Distinctive Regional Differences: a Cross-sectional Study
Status: Completed | Type: Observational
Sponsor: Sindh Institute of Urology and Transplantation (Other)
Responsible Party: Principal Investigator, Murk Niaz, Medical Officer, Sindh Institute of Urology and Transplantation
Other Study IDs: Breast Audit
Record Dates: First submitted 2022-07-14; First posted 2022-07-18 (Actual); Last update posted 2022-07-21 (Actual); Status verified 2022-07

CONDITIONS: Breast Cancer; Breast Neoplasms; Breast Cancer Invasive; Breast Cancer Stage; Breast Cancer Metastatic
Keywords: Breast cancer; Clinical audit; Breast cancer risk factors; Breast cancer screening; Clinicopathological characterisitics
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with breast cancer

SUMMARY:
This cross-sectional study, conducted at the Sindh Institute of Urology and Transplantation (SIUT), involved a retrospective data review of all the patients diagnosed with breast cancer from March 2017 to December 2021. The demographic characteristics, clinical presentation, stage of the disease, and histopathological characteristics were analyzed.

ELIGIBILITY:
Inclusion Criteria:

* All patients diagnosed with breast cancer

Exclusion Criteria:

* The patients that were lost to follow-up after the first consultation and those consulting for a second opinion were excluded from the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All breast cancer patients registered at the Breast Clinic, at the Sindh Institute of Urology and Transplantation (SIUT), Karachi from March 2017 till December 2021 were included
Sampling Method: Non-Probability Sample
Enrollment: 690 (Actual)
Dates: Start 2022-02-28 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
Demographic characteristics of patients with breast cancer | At the time of presentation
  age, gender, residence, marital status
Risk factors of patients with breast cancer | At the time of presentation
  age at menarche, menopause, parity, breastfeeding, contraception, family history, body mass index
Clinical presentation of patients with breast cancer | At the time of presentation
  site and duration
Stage of the breast cancer | At the time of presentation
  American Joint Committee on Cancer (AJCC) Anatomic Stage Groups for breast cancer
Histopathological characteristics of patients with breast cancer | At the time of presentation
  tumor type, hormone receptor status, Ki-67, and grade

CONTACTS AND LOCATIONS:
Overall Officials: Murk Niaz, Principal Investigator — Sindh Institute of Urology and Transplantation; Bushra Shirazi, Principal Investigator — Sindh Institute of Urology and Transplantation
Locations (1):
- Sindh Institute of Urology and Transplantation, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No